CLINICAL TRIAL: NCT05515484
Title: Improvement of Lung and Thoracic Compliance in ARDS Patients in Prone Position by Using Inflatable Air Bag
Acronym: MAPIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0195
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: ARDS; Prone Position; Mechanical Ventilation; Airbag
Keywords: ARDS; prone position; mechanical ventilation; airbag
MeSH Terms: interventions — Prone Position; Air Bags

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prone position with airbags (Experimental)
  Interventions: Other: prone position with airbags
- prone position standard of care (Active Comparator)
  Interventions: Other: prone position without airbags

INTERVENTIONS:
Other: prone position with airbags — prone position with airbags
  Arms: Prone position with airbags
Other: prone position without airbags — prone position without airbags
  Arms: prone position standard of care

SUMMARY:
ARDS is frequent in ICU and may lead to many complications and to death. Prone position is widely used in ADRS patients and demonstrated to decrease mortality. Regarding the chest wall compliance data are missing but the theorical response is that this compliance is decreased in a prone position mainly due to anterior chest and abdomen compression in this position which are more compliant that dorsal part of the body. As well prone position could be associated with complications as pressure ulcers. Because prone position is associated with complications, air bag were developped to decrease pressure on the chest and abdomen and to decrease pressure ulcers. Then, trying to improve chest compliance in prone position and reducing the risk of pressures ulcers could be a challenge with this system in comparison with standard care.

ELIGIBILITY:
Inclusion Criteria:

* patients with ARDS under mechanical ventilation with P/F ratio<150
* Age >18 y/o
* Admitted in the medical ICU of Amiens under mechanical ventilation sedated,
* With signed informed consent (patient or relative if patient is not conscious)

Exclusion Criteria:

* patients not eligible for a prone position
* Patients with tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
variation of Lung compliance between both groups | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No